CLINICAL TRIAL: NCT02117271
Title: "BEAUTY CPAP": The Impact of the Treatment of Obstructive Sleep Apnea With Continuous Positive Airway Pressure on Appearance and Age: a Randomized Crossover Placebo-controlled Study
Brief Title: The Treatment of Obstructive Sleep Apnea With Continuous Positive Airway Pressure on Appearance and Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nucleo Interdisciplinar da Ciencia do Sono (Other)
Responsible Party: Principal Investigator, Geraldo Lorenzi Filho, MD, PhD, Nucleo Interdisciplinar da Ciencia do Sono
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0068
Record Dates: First submitted 2014-04-10; First posted 2014-04-17 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; treatment; placebo; appearance; skin quality
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nasal dilator strip (Placebo Comparator): Breathe Right ® nasal dilator strip used during sleep
  Interventions: Other: Breathe Right ®
- continuous positive airway pressure (Experimental): nasal continuous positive airway pressure used during sleep
  Interventions: Device: continuous positive airway pressure

INTERVENTIONS:
Device: continuous positive airway pressure — device to treat obstructive sleep apnea using positive airway pressure with a nasal mask
  Other Names: Philips Respironics, System One, REMstar Pro
  Arms: continuous positive airway pressure
Other: Breathe Right ® — Nasal dilator strip treatment used during sleep to open the nasal airway
  Other Names: GlaxoSmithKline Brasil Ltda.
  Arms: nasal dilator strip

SUMMARY:
The investigators hypothesized that the treatment of obstructive sleep apnea (OSA) with continuous positive airway pressure (CPAP) will positively affect the appearance of the patient. The purpose of this study was to compare effects of one month of treatment of CPAP and placebo on appearance of patient with OSA in a randomized and crossover study.

Consecutive sleepy patients with severe OSA were included. The patients underwent three polysomnograms (PSG): first one to confirm OSA and two additional ones using placebo (nasal dilator) and for CPAP titration before starting each treatment period. All patients were randomly included into two treatment groups: 1) placebo use and 2) CPAP use. After one month with the first treatment and 15 days of washout, patients were crossed-over for the second treatment. Photographs from the patients' faces were obtained in the three experimental moments. The photographs were presented in a random order by the Qualtrics Survey Software, and were evaluated online by 704 observers for quantifying healthy appearance (unhealthy to extremely healthy), attractive (unattractive to extremely attractive) and tired (not tired to extremely tired). Apparent age was also rated for each observer. Quantitative evaluations of the skin characteristics of the patients' faces were also carried out at each experimental moment, including the presence of acne, patches, porosity, wrinkles, texture, and skin tone uniformity, through the capture of images by VISIATM System equipment.

During treatment period, the 30 patients (age = 46±9 years, 21 men) wearing placebo intervention on 98% of the nights and adherence to CPAP was 94%, with a mean of 6.0 ± 1.7 hours of use per day of treatment. Observational assessment of the photographs showed that patients were evaluated as being younger after using CPAP (P <0.001), but no quantitative changes in face skin characteristics were observed compared to the baseline and after the use of placebo.

Sleepy patients with severe OSA had a younger appearance after one month of CPAP treatment.

DETAILED DESCRIPTION:
Introduction: A previous study showed that sleep deprived people were perceived as less healthy, less attractive, and more tired than after a normal night's sleep (Axelsson et al., Beauty sleep: experimental study on the perceived health and attractiveness of sleep deprived people. BMJ 2010;341:c6614). The investigators believe that likewise sleep deprivation, patients with OSA also are perceived as less attractive, tired, healthy and look older than your age. the investigators therefore hypothesized that the treatment of OSA with continuous positive airway pressure (CPAP) positively affect the appearance of the patient. The purpose of this study was to compare effects of one month of treatment of CPAP and placebo on appearance of patient with OSA in a randomized and crossover study.

Methods:The investigators included 30 consecutive patients of both genders, aged between 30 and 60 years, referred to the sleep clinic of the Heart Institute (InCor) of University of Sao Paulo, with a history of snoring, excessive sleepiness, and with severe OSA confirmed by polysomnography. Patients were excluded if presenting previous treatment for sleep-disordered breathing, previous diagnosis of chronic diseases that interfere with sleep patterns and history the chronic use of alcohol, sedatives or drugs of abuse, in the last month.

Patients were randomized into two treatment groups: 1) Placebo arm - use of nasal dilator strip; and 2) CPAP arm - use of CPAP. At the first night of each treatment the patients were submitted to a polysomnography with nasal strip (placebo arm) or to CPAP titration (CPAP arm). After one month of treatment in the first randomized arm, patients were submitted to two weeks without treatment (washout period). After washout period, patients were assigned to the treatment crossover, i.e., patients in group 1) receiving CPAP therapy and patients in Group 2) receiving placebo treatment, during a period of one additional month. Excessive sleepiness (Epworth Sleepiness Scale) and quality of life (Functional Outcomes of Sleep Questionnaire - FOSQ) were evaluated in the three experimental times: baseline (immediately before treatment), one month (after one month of treatment defined at baseline), and 2 months (after one month of treatment crossover).

During the study period, the patients were followed by trained professionals and received all the necessary information about the use of each treatment. After three days of treatment, patients were contacted by phone to ensure the adherence treatment and to solve potential doubts. After each week of treatment, patients returned to the sleep clinic to management of the adherence data from the memory card (CPAP group) and data from the full filled sleep log (Placebo group), and also to had reinforced the information about the study protocol. Any issues or concerns about the treatment were also solved by phone calls.

All patients were photographed in the three experimental times: baseline (immediately before treatment), one month (after one month of treatment defined at baseline) and 2 months (after one month of treatment crossover). Photographs were taken by a trained photographer in a standardized manner. The photographer was blind to the experimental condition of patients. The photographs were displayed in a randomized order for 704 observers (general population, both genders, similar socioeconomic status and education), who were unaware of the conditions of the study. The observers rated the faces for attractiveness (very unattractive to very attractive), health (very sick to very healthy), and tiredness (not at all tired to very tired). Perceived age was also rated by the observers' evaluation by the Qualtrics Survey Software.

The high-resolution analyzing system VISIA TM (Canfield Scientific Inc. Fairfield USA) was used for computer analysis to precisely measure presence of porphyrins (P. acnes), coloration/evenness, vascular features, porosity, wrinkles and skin texture of the patient's face. The photographs from VISIA TM were taken after standard skin preparation and were analyzed by a specific analysis algorithm. Collection of dermatological assessments was conducted in three experimental sampling times.

During treatment period, the patients wearing placebo intervention on 98% of the nights and adherence to CPAP was 94%, with a mean of 6.0 ± 1.7 hours of use per day of treatment. After CPAP treatment, compared to baseline and after placebo treatment, improvement in the objective sleep quality, sleepiness, quality of life and depressive symptoms were observed (P <0.05). Observational assessment of the photographs showed that patients were evaluated as being younger after using CPAP (P <0.001), but no quantitative changes in face skin characteristics were observed compared to the baseline and after the use of placebo. Linear regression analysis identified the number of days with CPAP treatment, total sleep time and percentage of total sleep time with oxyhemoglobin saturation below 90% were predictors of decreasing of rated age after CPAP treatment.

In conclusion, sleepy patients with severe OSA had a younger appearance after one month of CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* severe sleep apnea (apnea-hypopnea index > 30)
* Epworth Sleepiness Scale score > 10

Exclusion Criteria:

* previous treatment for sleep-disordered breathing
* previous diagnosis of chronic diseases that interfere with sleep patterns
* history the chronic use of alcohol, sedatives or drugs of abuse, in the last month.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
appearance | 1 month
  Patients will be rated for attractiveness (very unattractive to very attractive), health (very sick to very healthy), tiredness (not at all tired to very tired) and age

SECONDARY OUTCOMES:
skin quality | 1 month
  Computer analysis of face image to measure presence of porphyrins (P. acnes), coloration/evenness, vascular features, porosity, wrinkles and skin texture.

CONTACTS AND LOCATIONS:
Overall Officials: GERALDO L FILHO, MD, PHD, Principal Investigator — University of Sao Paulo
Locations (1):
- Nucleo Interdisciplinar Da Ciencia Do Sono, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Yagihara F, Lorenzi-Filho G, Santos-Silva R. Patients With OSA Are Perceived as Younger Following Treatment With CPAP. Chest. 2019 Sep;156(3):553-561. doi: 10.1016/j.chest.2019.03.015. Epub 2019 Mar 27. PMID 30926396